CLINICAL TRIAL: NCT01035528
Title: Healthy Heart Study: Can Insulin Glargine Improve Myocardial Function in Patients With Type 2 Diabetes and Coronary Artery Disease? A Prospective, Randomized, Controlled Clinical Study With Blinded Analysis of Ultrasound Data
Brief Title: Can Insulin Glargine Improve Myocardial Function in Patients With T2D and Coronary Artery Disease (CAD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Munich Municipal Hospital (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Prof. Dr. Helene von Bibra, Munich Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HealthyHeart; HOE 901/6035 (Other: Aventis-Sanofi)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2004-08

CONDITIONS: Coronary Artery Disease; Type 2 Diabetes
Keywords: diastolic function, postmeal glucose, insulin glargine
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin glargine (Active Comparator): antidiabetic treatment with Lantus o.d. titrated to the target fasting glucose type 2 diabetes ≤110 mg/dl
  Interventions: Drug: insulin glargine
- metformin (Active Comparator): use of oral metformin o.d or b.d titrated up to 2000 mg daily for to the target fasting glucose ≤110 mg/dl
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: insulin glargine — antidiabetic treatment with insulin glargine sc o.d. titrated to the target fasting glucose type 2 diabetes ≤110 mg/dl
  Other Names: Lantus
  Arms: insulin glargine
Drug: metformin — use of oral metformin o.d or b.d titrated up to 2000 mg daily for to the target fasting glucose ≤110 mg/dl
  Other Names: Siofor
  Arms: metformin

SUMMARY:
The field of secondary prevention remains an extremely important goal for diagnostic and therapeutic approaches keeping in mind that 40% of all patients with acute myocardial infarction have prediabetes, commonly as impaired glucose tolerance, which has not been known and treated and for which there are no guidelines for treatment. In this context, accumulating evidence shows beneficial effects for treating diabetes mellitus early in the course of disease, whereas other evidence shows that aggressive antidiabetic therapy may be associated with undesired risks. Accordingly, the present randomized and controlled pilot study is designed as hypothesis creating study to create first data about potential medication in early type 2 diabetes including impaired glucose tolerance of patients with known coronary artery disease as means of secondary prevention by comparing oral antidiabetic therapy with metformin with insulin glargine o.d. and by studying the respective effects on cardiovascular function and metabolism both in the fasting state and after a standardized meal. As diastolic myocardial function has emerged as important prognosticator, the hypothesis was tested that treatment with insulin glargine improves myocardial function in patients with coronary artery disease and newly diagnosed type 2 diabetes including impaired glucose tolerance.

DETAILED DESCRIPTION:
This is a single centre, short term (24 weeks), therapy controlled and randomized prospective study with blinded analysis of the ultrasound data in 28 patients with known coronary artery disease, normal systolic cardiac function and with newly diagnosed type 2 diabetes including impaired glucose tolerance who are treated by ≤1 oral antidiabetic medication. After recruitment and informed consent, patients are randomized to two treatment arms which takes into account age and presence or absence of therapy with statins.

In one treatment arm, therapy is based on insulin glargine sc o.d., while in the other treatment arm, therapy is based on oral metformin, up to 2000 mg daily. Both treatment arms will be titrated to the target of fasting glucose ≤110 mg/dl during the first 12 weeks. The patients in the insulin treatment arm will be instructed in the skills of self-medication by the departmental diabetic teaching programme prior to starting study medication and are encouraged to keep records of any episode of hypoglycemia throughout the study.Outpatients visits for metabolic control and ultrasound assessment are at weeks 4, 12 and 24 after baseline and are associated with life style instructions for all patients.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease
* type 2 diabetes of short duration including impaired glucose tolerance and impaired fasting glucose
* treatment by ≤1 OAD

Exclusion Criteria:

* contraindications for metformin or insulin glargine
* on insulin therapy
* pregnancy and breastfeeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2005-04; Primary Completion 2010-02 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
change from baseline to endpoint in myocardial diastolic velocity E' | 24 weeks

SECONDARY OUTCOMES:
glucose control | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helene von Bibra, MD, PhD, Principal Investigator — Diabetes Centre, Staedt. Klinikum Bogenhausen, Muenchen
Locations (1):
- Staedt. Klinikum Muenchen Bogenhausen, Munich, Bavaria, Germany